CLINICAL TRIAL: NCT00231530
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Safety and Efficacy of Topiramate in the Treatment of Obese, Type 2 Diabetic Patients on a Controlled Diet
Brief Title: A Study of the Safety and Efficacy of Topiramate in the Treatment of Obese, Type 2 Diabetes Patients on a Controlled Diet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003712
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus, Adult-Onset
Keywords: Type 2 Diabetes Mellitus; Obesity; Diabetic Diet; Hypertension; Hyperlipidemia; Adult-Onset Diabetes Mellitus(AODM)
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Hypertension; Hyperlipidemias | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to determine the efficacy and safety of topiramate compared with placebo in obese, Type 2 diabetic patients on a controlled diet.

DETAILED DESCRIPTION:
Topiramate is not approved for the treatment of obesity. This is a randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of topiramate in obese, diet-controlled, type 2 diabetic patients. Patients are randomized to receive either topiramate or placebo. After a 5 week pre-enrollment phase followed by a 6 week run-in phase, patients in the topiramate group start an 8-week titration phase to reach the assigned dose of topiramate, either 96 or 192 mg daily. Treatment continues for 1 year. Assessments of effectiveness include percent change in body weight, hemoglobin type A1c [HbA1c] levels, Body Mass Index [BMI], the numbers and proportion of 5% and 10% weight loss responders, glucose tolerance, waist and hip circumferences, changes in the mass of left ventricle of the heart, blood pressures, and fasting lipid profiles. Safety evaluations, including incidence of adverse events, vital signs, clinical laboratory values, and electrocardiograms [ECGs], are monitored throughout the study. The study hypothesis is that topiramate, combined with controlled diet, will be effective in weight reduction and controlling blood sugar level and is well tolerated. During the initial 8 weeks, the oral doses of either a matching placebo or topiramate will be gradually increased to the target doses (96 milligrams[mg] or 192mg daily); the dose will be maintained for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index >= 27 and < 50
* Diagnosis of Type 2 diabetes according to either Swedish guideline or the American Diabetes Association (ADA) criteria
* HbA1c <10.5% at enrollment
* No previous oral antidiabetic medication or insulin therapy
* Stable body weight
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing an acceptable method of contraception (requires negative pregnancy test)

Exclusion Criteria:

* Known contraindication or hypersensitivity to topiramate
* Fasting plasma glucose (FPG) >= 13.1 millimolesl/liter (240 milligrams/deciliter) at baseline, Visit 4 (Week 0)
* HBA1c of >10.5% at enrollment
* History of severe recurrent hypoglycemic episodes prior to study entry
* Use of any systemic corticosteroids within 30 days of enrollment
* Diagnosed Type 1 diabetes
* History of significant cardiovascular disease, uncontrolled thyroid disease, or kidney stones

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2001-01; Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
The percent change in body weight and change in Hemoglobin A1c from enrollment to Week 60.

SECONDARY OUTCOMES:
Change from enrollment or baseline to Week 60 in BMI, waist circumference, glucose tolerance, lipid profile; safety measures, such as adverse events, throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Study of the Safety and Efficacy of Topiramate in the Treatment of Obese, Type 2 Diabetes Patients on a Controlled Diet — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=536&filename=CR003712_CSR.pdf